CLINICAL TRIAL: NCT06927063
Title: Long-term Recovery and Microbiota-Gut-Brain Axis Disruption After Traumatic Brain Injury
Acronym: OVERCOME-TBI
Status: Not yet recruiting | Type: Observational
Sponsor: Turku University Hospital (Other Government)
Collaborators: Aalto University (Other); University of Geneva, Switzerland (Other); Göteborg University (Other); University of Cambridge (Other); Örebro University, Sweden (Other); University of Turku (Other)
Responsible Party: Sponsor
Other Study IDs: 21/1801/2022; 21/1801/2022 (Other: Hospital District of Southwest Finland)
Record Dates: First submitted 2024-06-10; First posted 2025-04-15 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Traumatic Brain Injury
Keywords: traumatic; brain; injury; traumatic brain injury; TBI; neuroinflammation; gut; microbiota; microbiota-gut-brain axis; DTI; diffusion tensor; biomarker; blood based biomarker
MeSH Terms: conditions — Brain Injuries, Traumatic; Wounds and Injuries; Neuroinflammatory Diseases | interventions — Diffusion Magnetic Resonance Imaging; Positron-Emission Tomography

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 14 Years
Biospecimen Retention: Samples With DNA — blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with history of sustained traumatic brain injury: Patients with history of sustained traumatic brain injury 1-4 and 11-14 years earlier
  Interventions: Diagnostic Test: blood-based protein biomarker assessments; Diagnostic Test: blood-based metabolomic/lipidomic biomarker assessments; Diagnostic Test: Diffusion-weighted magnetic resonance imaging (brain); Diagnostic Test: Structural magnetic resonance imaging (brain); Diagnostic Test: PET imaging (brain); Procedure: Standard colonoscopy with pinch biopsies; Diagnostic Test: Fecal microbiome assessments
- Control patients with history of orthopedic injury without traumatic brain injury: Patients with history of sustained orthopedic injury without traumatic brain injury 1-4 and 11-14 years earlier
  Interventions: Diagnostic Test: blood-based protein biomarker assessments; Diagnostic Test: blood-based metabolomic/lipidomic biomarker assessments; Diagnostic Test: Diffusion-weighted magnetic resonance imaging (brain); Diagnostic Test: Structural magnetic resonance imaging (brain); Diagnostic Test: PET imaging (brain); Procedure: Standard colonoscopy with pinch biopsies; Diagnostic Test: Fecal microbiome assessments

INTERVENTIONS:
Diagnostic Test: blood-based protein biomarker assessments — Assessment of multiple blood-based biomarkers of different cellular origin and inflammatory mediators
Diagnostic Test: blood-based metabolomic/lipidomic biomarker assessments — Assessment of multiple blood-based TBI-related metabolomic and lipidomic biomarkers
Diagnostic Test: Diffusion-weighted magnetic resonance imaging (brain) — Diffusion-weighted magnetic resonance imaging
Diagnostic Test: Structural magnetic resonance imaging (brain) — Structural magnetic resonance imaging
Diagnostic Test: PET imaging (brain) — Positron emission tomography imaging
Procedure: Standard colonoscopy with pinch biopsies — Standard colonoscopy including pinch biopsies from the bowel wall at several levels (terminal ileum, ascending colon, transverse colon, descending colon, and rectosigmoideum) for histology, microbiome analysis and metabolomics
Diagnostic Test: Fecal microbiome assessments — Fecal microbiome assessments (DNA)

SUMMARY:
The OVERCOME-TBI project aims to collect multimodal data approximately 1-4 and 11-14 years after an earlier well-documented traumatic brain injury (TBI) and examine factors that influence disease progression in order to gain new scientific insights into the long-term pathophysiology of TBI and identify new therapeutic targets.

TBIs are among the most serious health problems worldwide and represents a significant burden for the injured, their families and society. It is estimated that more than 50 million people in the world suffer a TBI every year and half of all people will suffer a TBI in their lifetime. TBI diagnostics has lagged significantly behind that of many other diseases. The current methods for assessing severity and predicting outcomes are based only on initial stage variables, and there are no objective tools for monitoring disease progression. The current acute severity indices have shown only a modest association with outcome, particularly in patients with mTBI. However, even in patients with moderate-severe TBI, clinical predictors and imaging together explain only 35% of the variance in outcomes.

In the OVERCOME-TBI project, patients with a history of TBI sustained 1-4 and 11-14 years earlier will undergo extensive neurological, biochemical, microbiological, gastroenterological and imaging examinations. The patients have previously participated in the prospective studies of our research group, so that data on acute injuries, blood-based biomarkers and advanced imaging results are already available. The results are expected to yield objective diagnostic and treatment methods for the diagnosis of progressive brain disease after brain injury and for the identification of microbiome-gut-brain axis dysfunction associated with disease progression.

DETAILED DESCRIPTION:
This detailed description outlines the scientific background, registry procedures and quality control strategies for the OVERCOME-TBI study. The study builds on previous research cohorts Evidence-based Diagnostic and Treatment Planning Solution for Traumatic Brain Injuries) and PACoS-TBI (Pathophysiological Characterization of Severe Traumatic Brain Injury) and aims to comprehensively investigate long-term outcomes and the role of the microbiome-gut-brain axis in traumatic brain injury (TBI) through multimodal and longitudinal and cross-sectional data collection.

The OVERCOME-TBI study uses a prospective observational design focusing on patients with moderate and severe TBI. It includes both recently injured TBI patients and long-term survivors to capture a broad trajectory of recovery from TBI. The study will include a broad range of modalities, including clinical assessments, neurocognitive testing, advanced neuroimaging (MRI, PET-MRI), blood biomarkers, microbiome analysis and optional endoscopic biopsies. This integrated approach is structured to provide insights into complex biological mechanisms that influence TBI outcomes.

The overall goal of the OVERCOME-TBI project is to collect multimodal data approximately 1-4 and 11-14 years after a previous, well-documented TBI and to investigate factors that influence disease progression in order to gain new scientific insights into the long-term pathophysiology of TBI and to identify new therapeutic targets. The core of the study design involves the prior collection of extensive clinical, radiological and molecular data at multiple time points: acute hospitalization (0-7 days post-injury), early follow-up (3-6 months) and long-term follow-up (≥12 months). Clinical outcomes are assessed using validated instruments such as the Glasgow Outcome Scale - Extended (GOSE) and the Rivermead Post-Concussion Symptoms Questionnaire (RPQ). These assessments aim to capture both functional and cognitive recovery patterns. The other part of the data collection includes cross-sectional data 1-4 and 11-14 years after TBI.

In terms of registry procedures, each participant is documented in a comprehensive electronic case report form (CRF) that includes demographic information, injury details, ICU and hospital course, surgical interventions, and rehabilitation history. CRFs are created and maintained electronically via secure hospital systems. All CRFs are protected by user authentication. The registry also includes a register of study participants that is created and maintained in accordance with EU General Data Protection Regulation (GDPR) guidelines to ensure participant confidentiality and regulatory compliance.

The biological component of the study includes the collection and storage of peripheral blood, stool samples and, if possible, intestinal biopsies. The blood is collected at predefined intervals and processed into serum and plasma. These are stored at -70°C under biobank conditions with standardized protocols to ensure consistency. Stool samples are taken for microbiome analysis and biopsies, if performed, are stored at -70°C. All samples are pseudonymized and tracked using unique identifiers.

Sample analyzes are performed in several specialized laboratories, including the University of Turku (Finland), the University of Geneva (Switzerland), Sahlgrenska University Hospital (Sweden), and Örebro University (Sweden). Standard operating procedures (SOPs) were developed for blood biomarker assays, microbiome profiling and inflammatory cytokine analysis. Cross-laboratory calibration and quality control measures are instituted to ensure reproducibility and cross-site comparability.

The neuroimaging component includes MRI and PET-MRI. MRI sequences include T1-weighted, FLAIR, SWI and DTI to assess structural and microstructural changes. PET imaging is performed with radioligands that target translocator protein (TSPO) expression and provide insight into neuroinflammation. Imaging data will be analyzed centrally in Turku and Cambridge using harmonized pipelines and machine learning based segmentation methods.

Functional and cognitive assessments are an integral part of the protocol. In addition to GOSE and RPQ, the CANTAB test battery is performed. These tests aim to identify common neuropsychiatric sequelae and investigate correlations with biological and imaging markers.

Data protection and management procedures are a central part of the protocol. All data collected will be entered into a secure, GDPR-compliant data platform. Anonymization is achieved through pseudonymization and encryption strategies. A data access committee regulates data sharing and all shared datasets are derived from anonymized master files as part of data usage agreements. The central database is hosted at Turku University Hospital and is subject to strict backup and archiving protocols.

Informed consent will be obtained from all participants or their legal representatives prior to inclusion in the study. The procedure includes an oral explanation, a written information sheet and time for questions. For cognitively impaired patients, a proxy consent will be documented according to the guidelines of the local ethics committee. All consent forms will be kept in the participant's CRF.

The study has been approved by the Ethics Committee of the Wellbeing Services County of Southwest Finland and the Clinical Services of the Wellbeing Services County of Southwest Finland complies with the Declaration of Helsinki. Procedures involving radiation (PET-MRI) and invasive sampling (biopsy) will be performed within established safety limits. Risk management protocols identify potential harm and define measures for adverse events.

Quality control is embedded in every phase of the study. Standardization of data collection, harmonization of sample handling, staff training and audit trails for all data entries are emphasized.

To address potential sample size limitations or data heterogeneity, the protocol includes provisions for external collaboration. In particular, the study is aligned with the international InTBIR (International Initiative for Traumatic Brain Injury Research) framework, which facilitates data pooling and harmonization with global datasets.

Analysis strategies include logistic regression, linear mixed models and machine learning classifiers. Multimodal fusion analyzes will examine associations between neuroimaging features, cognitive outcomes and biological markers. Time series data will be used to identify trajectories and phenotypes of recovery. Missing data will be treated with multiple imputation or maximum likelihood methods with complete information, depending on the analysis.

Documentation and archiving are performed according to international standards. All physical documentation will be stored securely and electronic files will be stored on institutional servers with restricted access. Research data is retained for at least 20 years.

The study is funded by the Research Council of Finland, the Sigrid Jusélius Foundation and the Finnish State Research Funding. Insurance coverage is provided by Turku University Hospital and covers all patient-related research activities.

In summary, the OVERCOME-TBI protocol represents a comprehensive, ethically sound and scientifically rigorous study framework. It integrates high-quality registry methods, biological sample analysis, cognitive and gastrointestinal assessments, and state-of-the-art imaging. Quality assurance is enforced through robust procedures at all levels to achieve reliable, generalizable and clinically meaningful results in the field of TBI research.

ELIGIBILITY:
Inclusion Criteria:

* All those who are alive and give their consent will be included from our previous prospective studies (TBIcare or PACoS-TBI)

Exclusion Criteria (neurological and imaging studies):

* For patients with TBI there are no exclusion criteria, and all eligible patients who give consent will be recruited
* Those patients and controls with contraindication for head MRI (MRI-incompatible heart pacemaker, weight over 200 kg, mechanical heart valve prosthesis, first trimester of pregnancy, orbital area tattoo) will not undergo head MRI. Instead, they we will undergo the other assessments
* For controls, those who have suffered a TBI or any other brain disorder after the TBIcare or PACoS-TBI study will be excluded.

Exclusion Criteria (colonoscopy)

* Diagnosis of IBD or other diagnosis besides IBS causing severe GI symptoms, such as microscopic colitis or bile acid diarrhea
* Poorly controlled celiac disease
* Colorectal cancer diagnosed within five years
* Antibiotic or probiotic treatment, on-going or previous month.
* Unwilling or unable to undergo colonoscopy and/or standard bowel preparation.
* Significantly increased risk of heart or kidney failure or electrolyte imbalances due to bowel preparation (frailty, serious pre-existing heart or kidney insufficiency).
* Altered bowel anatomy after significant operation. Appendicectomy or cholecystectomy are considered minor operations.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All those who are alive and give their consent will be included from our previous prospective studies (TBIcare or PACoS-TBI)
Sampling Method: Non-Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Biochemical neuroinflammation burden (lipids and metabolites) | 1-14 years after traumatic brain injury
  Neuroinflammation burden as measured by levels of blood-based lipid biomarkers choline phospholipids (lysophosphatidylcholines, ether phosphatidylcholines, and sphingomyelins), branched-chain amino acids and medium-chain fatty acids
Biochemical neuroinflammation burden (cytokines) | 1-14 years after traumatic brain injury
  Neuroinflammation burden as measured by levels of blood-based cytokines IL-6, IL-15, and MCP-1
Functional outcome | 1-14 years after traumatic brain injury
  Functional outcome measured with Glasgow Outcome Scale Extended (GOSE, 1=dead - 8=complete recovery)
Changes in microbiota | 1-14 years after traumatic brain injury
  DNA from fecal microbiome assessed by deep shot gun metagenomics approach, referenced to a population of healthy control subjects
Inflammation burden on head positron emission tomography | 1-14 years after traumatic brain injury
  Neuroinflammation measured using the [11C]PK11195 radioligand

SECONDARY OUTCOMES:
Changes in brain white and grey matter microstructure | 1-14 years after traumatic brain injury
  Changes in brain white and grey matter microstructure as measured with diffusion tensor metrics
Accelerated brain ageing | 1-14 years after traumatic brain injury
  Accelerated brain ageing calculated at a whole brain level using T1-weighted images and at a voxel-based level as the annualised Jacobian determinants in white matter and grey matter, referenced to a population of healthy control subjects

CONTACTS AND LOCATIONS:
Overall Officials: Jussi P. Posti, MD, PhD, Principal Investigator — Turku University Hospital and University of Turku

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Newcombe VFJ, Ashton NJ, Posti JP, Glocker B, Manktelow A, Chatfield DA, Winzeck S, Needham E, Correia MM, Williams GB, Simren J, Takala RSK, Katila AJ, Maanpaa HR, Tallus J, Frantzen J, Blennow K, Tenovuo O, Zetterberg H, Menon DK. Post-acute blood biomarkers and disease progression in traumatic brain injury. Brain. 2022 Jun 30;145(6):2064-2076. doi: 10.1093/brain/awac126. PMID 35377407
- [Result] Shahim P, Politis A, van der Merwe A, Moore B, Ekanayake V, Lippa SM, Chou YY, Pham DL, Butman JA, Diaz-Arrastia R, Zetterberg H, Blennow K, Gill JM, Brody DL, Chan L. Time course and diagnostic utility of NfL, tau, GFAP, and UCH-L1 in subacute and chronic TBI. Neurology. 2020 Aug 11;95(6):e623-e636. doi: 10.1212/WNL.0000000000009985. Epub 2020 Jul 8. PMID 32641529
- [Result] Sundman MH, Chen NK, Subbian V, Chou YH. The bidirectional gut-brain-microbiota axis as a potential nexus between traumatic brain injury, inflammation, and disease. Brain Behav Immun. 2017 Nov;66:31-44. doi: 10.1016/j.bbi.2017.05.009. Epub 2017 May 17. PMID 28526435
- [Result] Patterson TT, Nicholson S, Wallace D, Hawryluk GWJ, Grandhi R. Complex Feed-Forward and Feedback Mechanisms Underlie the Relationship Between Traumatic Brain Injury and the Gut-Microbiota-Brain Axis. Shock. 2019 Sep;52(3):318-325. doi: 10.1097/SHK.0000000000001278. PMID 30335675
- [Result] undefined
- [Result] Cryan JF, Dinan TG. Mind-altering microorganisms: the impact of the gut microbiota on brain and behaviour. Nat Rev Neurosci. 2012 Oct;13(10):701-12. doi: 10.1038/nrn3346. Epub 2012 Sep 12. PMID 22968153
- [Result] Dinan TG, Cryan JF. The impact of gut microbiota on brain and behaviour: implications for psychiatry. Curr Opin Clin Nutr Metab Care. 2015 Nov;18(6):552-8. doi: 10.1097/MCO.0000000000000221. PMID 26372511
- [Result] Jassam YN, Izzy S, Whalen M, McGavern DB, El Khoury J. Neuroimmunology of Traumatic Brain Injury: Time for a Paradigm Shift. Neuron. 2017 Sep 13;95(6):1246-1265. doi: 10.1016/j.neuron.2017.07.010. PMID 28910616
- [Result] Koerte IK, Lin AP, Muehlmann M, Merugumala S, Liao H, Starr T, Kaufmann D, Mayinger M, Steffinger D, Fisch B, Karch S, Heinen F, Ertl-Wagner B, Reiser M, Stern RA, Zafonte R, Shenton ME. Altered Neurochemistry in Former Professional Soccer Players without a History of Concussion. J Neurotrauma. 2015 Sep 1;32(17):1287-93. doi: 10.1089/neu.2014.3715. Epub 2015 May 14. PMID 25843317
- [Result] Coughlin JM, Wang Y, Munro CA, Ma S, Yue C, Chen S, Airan R, Kim PK, Adams AV, Garcia C, Higgs C, Sair HI, Sawa A, Smith G, Lyketsos CG, Caffo B, Kassiou M, Guilarte TR, Pomper MG. Neuroinflammation and brain atrophy in former NFL players: An in vivo multimodal imaging pilot study. Neurobiol Dis. 2015 Feb;74:58-65. doi: 10.1016/j.nbd.2014.10.019. Epub 2014 Nov 7. PMID 25447235
- [Result] Wilson L, Stewart W, Dams-O'Connor K, Diaz-Arrastia R, Horton L, Menon DK, Polinder S. The chronic and evolving neurological consequences of traumatic brain injury. Lancet Neurol. 2017 Oct;16(10):813-825. doi: 10.1016/S1474-4422(17)30279-X. Epub 2017 Sep 12. PMID 28920887
- [Result] Tenovuo O, Diaz-Arrastia R, Goldstein LE, Sharp DJ, van der Naalt J, Zasler ND. Assessing the Severity of Traumatic Brain Injury-Time for a Change? J Clin Med. 2021 Jan 4;10(1):148. doi: 10.3390/jcm10010148. PMID 33406786
- [Result] Posti JP, Dickens AM, Oresic M, Hyotylainen T, Tenovuo O. Metabolomics Profiling As a Diagnostic Tool in Severe Traumatic Brain Injury. Front Neurol. 2017 Aug 18;8:398. doi: 10.3389/fneur.2017.00398. eCollection 2017. PMID 28868043
- [Result] Mikolic A, Groeniger JO, Zeldovich M, Wilson L, van Lennep JR, van Klaveren D, Polinder S; Collaborative European NeuroTrauma Effectiveness Research in Traumatic Brain Injury (CENTER-TBI) Participants and Investigators. Explaining Outcome Differences between Men and Women following Mild Traumatic Brain Injury. J Neurotrauma. 2021 Dec;38(23):3315-3331. doi: 10.1089/neu.2021.0116. PMID 34617454
- [Result] Schneider ALC, Huie JR, Boscardin WJ, Nelson L, Barber JK, Yaffe K, Diaz-Arrastia R, Ferguson AR, Kramer J, Jain S, Temkin N, Yuh E, Manley GT, Gardner RC; TRACK-TBI Investigators. Cognitive Outcome 1 Year After Mild Traumatic Brain Injury: Results From the TRACK-TBI Study. Neurology. 2022 Mar 22;98(12):e1248-e1261. doi: 10.1212/WNL.0000000000200041. Epub 2022 Feb 16. PMID 35173018
- [Result] Nelson LD, Temkin NR, Dikmen S, Barber J, Giacino JT, Yuh E, Levin HS, McCrea MA, Stein MB, Mukherjee P, Okonkwo DO, Robertson CS, Diaz-Arrastia R, Manley GT; and the TRACK-TBI Investigators; Adeoye O, Badjatia N, Boase K, Bodien Y, Bullock MR, Chesnut R, Corrigan JD, Crawford K, Duhaime AC, Ellenbogen R, Feeser VR, Ferguson A, Foreman B, Gardner R, Gaudette E, Gonzalez L, Gopinath S, Gullapalli R, Hemphill JC, Hotz G, Jain S, Korley F, Kramer J, Kreitzer N, Lindsell C, Machamer J, Madden C, Martin A, McAllister T, Merchant R, Noel F, Palacios E, Perl D, Puccio A, Rabinowitz M, Rosand J, Sander A, Satris G, Schnyer D, Seabury S, Sherer M, Taylor S, Toga A, Valadka A, Vassar MJ, Vespa P, Wang K, Yue JK, Zafonte R. Recovery After Mild Traumatic Brain Injury in Patients Presenting to US Level I Trauma Centers: A Transforming Research and Clinical Knowledge in Traumatic Brain Injury (TRACK-TBI) Study. JAMA Neurol. 2019 Sep 1;76(9):1049-1059. doi: 10.1001/jamaneurol.2019.1313. PMID 31157856
- [Result] Brazinova A, Rehorcikova V, Taylor MS, Buckova V, Majdan M, Psota M, Peeters W, Feigin V, Theadom A, Holkovic L, Synnot A. Epidemiology of Traumatic Brain Injury in Europe: A Living Systematic Review. J Neurotrauma. 2021 May 15;38(10):1411-1440. doi: 10.1089/neu.2015.4126. Epub 2018 Dec 19. PMID 26537996
- [Result] Stewart WF, Kim N, Ifrah CS, Lipton RB, Bachrach TA, Zimmerman ME, Kim M, Lipton ML. Symptoms from repeated intentional and unintentional head impact in soccer players. Neurology. 2017 Feb 28;88(9):901-908. doi: 10.1212/WNL.0000000000003657. Epub 2017 Feb 1. PMID 28148633
- [Result] Priemer DS, Iacono D, Rhodes CH, Olsen CH, Perl DP. Chronic Traumatic Encephalopathy in the Brains of Military Personnel. N Engl J Med. 2022 Jun 9;386(23):2169-2177. doi: 10.1056/NEJMoa2203199. PMID 35675177
- [Result] Maas AIR, Menon DK, Manley GT, Abrams M, Akerlund C, Andelic N, Aries M, Bashford T, Bell MJ, Bodien YG, Brett BL, Buki A, Chesnut RM, Citerio G, Clark D, Clasby B, Cooper DJ, Czeiter E, Czosnyka M, Dams-O'Connor K, De Keyser V, Diaz-Arrastia R, Ercole A, van Essen TA, Falvey E, Ferguson AR, Figaji A, Fitzgerald M, Foreman B, Gantner D, Gao G, Giacino J, Gravesteijn B, Guiza F, Gupta D, Gurnell M, Haagsma JA, Hammond FM, Hawryluk G, Hutchinson P, van der Jagt M, Jain S, Jain S, Jiang JY, Kent H, Kolias A, Kompanje EJO, Lecky F, Lingsma HF, Maegele M, Majdan M, Markowitz A, McCrea M, Meyfroidt G, Mikolic A, Mondello S, Mukherjee P, Nelson D, Nelson LD, Newcombe V, Okonkwo D, Oresic M, Peul W, Pisica D, Polinder S, Ponsford J, Puybasset L, Raj R, Robba C, Roe C, Rosand J, Schueler P, Sharp DJ, Smielewski P, Stein MB, von Steinbuchel N, Stewart W, Steyerberg EW, Stocchetti N, Temkin N, Tenovuo O, Theadom A, Thomas I, Espin AT, Turgeon AF, Unterberg A, Van Praag D, van Veen E, Verheyden J, Vyvere TV, Wang KKW, Wiegers EJA, Williams WH, Wilson L, Wisniewski SR, Younsi A, Yue JK, Yuh EL, Zeiler FA, Zeldovich M, Zemek R; InTBIR Participants and Investigators. Traumatic brain injury: progress and challenges in prevention, clinical care, and research. Lancet Neurol. 2022 Nov;21(11):1004-1060. doi: 10.1016/S1474-4422(22)00309-X. Epub 2022 Sep 29. PMID 36183712
- [Result] Maas AIR, Menon DK, Adelson PD, Andelic N, Bell MJ, Belli A, Bragge P, Brazinova A, Buki A, Chesnut RM, Citerio G, Coburn M, Cooper DJ, Crowder AT, Czeiter E, Czosnyka M, Diaz-Arrastia R, Dreier JP, Duhaime AC, Ercole A, van Essen TA, Feigin VL, Gao G, Giacino J, Gonzalez-Lara LE, Gruen RL, Gupta D, Hartings JA, Hill S, Jiang JY, Ketharanathan N, Kompanje EJO, Lanyon L, Laureys S, Lecky F, Levin H, Lingsma HF, Maegele M, Majdan M, Manley G, Marsteller J, Mascia L, McFadyen C, Mondello S, Newcombe V, Palotie A, Parizel PM, Peul W, Piercy J, Polinder S, Puybasset L, Rasmussen TE, Rossaint R, Smielewski P, Soderberg J, Stanworth SJ, Stein MB, von Steinbuchel N, Stewart W, Steyerberg EW, Stocchetti N, Synnot A, Te Ao B, Tenovuo O, Theadom A, Tibboel D, Videtta W, Wang KKW, Williams WH, Wilson L, Yaffe K; InTBIR Participants and Investigators. Traumatic brain injury: integrated approaches to improve prevention, clinical care, and research. Lancet Neurol. 2017 Dec;16(12):987-1048. doi: 10.1016/S1474-4422(17)30371-X. Epub 2017 Nov 6. No abstract available. PMID 29122524

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-06-20): https://cdn.clinicaltrials.gov/large-docs/63/NCT06927063/Prot_SAP_000.pdf